CLINICAL TRIAL: NCT06261294
Title: CONQUER Cancer Study: To Collect Blood Samples From Cancer and Non-cancer Participants for Development and Validation of the 'OncoSweep Cancer Spotlight and Spectrum Product Line
Brief Title: OncoSweep Cancer Spotlight and Spectrum Product Line
Status: Completed | Type: Observational
Sponsor: Pharus Taiwan, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CPIP-LUN-A001
Record Dates: First submitted 2024-02-06; First posted 2024-02-15 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Lung Cancer
Keywords: cancer study
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- two group Study arm determination based: Subjects will be assigned into Test group or Control group based on the criteria:
  * Test group: Individual who has been diagnosed with lung nodule(s) or mass by his/ her healthcare provider utilizing LDCT or CT scan and has already scheduled for interventional procedure;
  * Control group: Individual is willing to undergo COPD examination and LDCT or CT scan with 3-5 mm spatial z-axis resolution and has no findings from the scan and examination
  Interventions: Diagnostic Test: OncoSweep Lung Spotligh

INTERVENTIONS:
Diagnostic Test: OncoSweep Lung Spotligh — This study is to develop and validate the performance of OncoSweep Lung Spotlight for detecting circulating miRNA expression, ctDNA methylation status, platelet RNA, and tumor marker expressions by utilizing real-time polymerase chain reaction (qPCR). The method is to collect venous blood from subjects during their routine visit to the healthcare facilities.

SUMMARY:
CONQUER cancer study: To collect blood samples from cancer and non-cancer participants for development and validation of the 'OncoSweep Cancer Spotlight and Spectrum Product Line'

DETAILED DESCRIPTION:
OncoSweep Cancer Spotlight and Spectrum Product Lines are qualitative in vitro diagnostic devices testing plasma specimens for detecting circulating miRNA expression, ctDNA methylation status, platelet RNA analysis, and tumor marker expressions by utilizing real-time polymerase chain reaction (qPCR) and next-generation sequencing (NGS). This is a two-arm, open-label, non-randomized controlled pilot study intends to screen adults 18 years or older, who are treatment-naïve for cancers and have pulmonary nodules or mass detected by low-dose computerized tomography (LDCT) or standard computerized tomography (CT) scans. OncoSweep Lung Spotlight will be utilized with venous blood samples collected in the healthcare facility where the study is being conducted. The X-ray, LDCT/ standard CT scan, blood laboratory test data, or biopsy results will be collected from the control group, and the blood sample will be analyzed by OncoSweep Lung Spotlight. Results generated from both groups will be evaluated against each other. The result of OncoSweep Lung Spotlight provides additional evidence to support or assist medical diagnoses when used in combination with LDCT/ standard CT scan data.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion

  1. Individual who is not mentally impaired, capable to read, understand, and is willing to provide signed and dated informed consent form.
  2. Individual is aged 18 years old or above.
  3. Individual who is willing to provide information on the given questionnaire. Test group: Individual was diagnosed with pulmonary nodules or masses by low-dose CT (LDCT)/ CT, and evaluated by the physician needed to conduct a biopsy or/ and surgery has been arranged.

     Control group: Individual is willing to undergo LDCT or CT scan with 3-5 mm spatial z-axis resolution, pulmonary function examination, X-ray, laboratory blood test, and blood drawing.
  4. Control group: Individual has no abnormal finding from LDCT or CT scan with 3-5 mm spatial z-axis resolution and pulmonary function examination(FEV1/FVC Ratio≧70%).
  5. Individual did not donate blood or receive blood transfusion within two months before joining the study.

Exclusion Criteria:

* Exclusion

  1. Individual who is not suitable for participating as per Investigator's judgement.
  2. Individual who has undergone gene therapy or related product within one year prior to enrolling in this study.
  3. Individual who is attending another clinical study at the time of enrollment.
  4. Individual who is known to be pregnant.
  5. Individual who has received a vaccine within two weeks.
  6. Individual who has a history of any cancer occurrences other than lung cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This is a two-arm, open-label, non-randomized controlled pilot study intended to screen adults of 18 years or older, who are treatment-naïve for cancers, or who have pulmonary nodules or masses detected by LDCT or standard CT scan, utilizing OncoSweep Lung Spotlight with venous blood sample collected in the healthcare facility where the study is being conducted.
Sampling Method: Non-Probability Sample
Enrollment: 109 (Actual)
Dates: Start 2023-05-29 (Actual); Primary Completion 2025-03-03 (Actual); Study Completion 2025-05-07 (Actual)

PRIMARY OUTCOMES:
To differentiate lung cancer signals from non-cancer signals based on analysis of OncoSweep Lung Spotlight. | two years
  To compare blood samples from lung cancer cases and non-cancer control subjects to develop and evaluate:1.Cancer models for discriminating lung cancer versus non-cancer 2.Platform evaluation 3.Data storage and algorithm establishment for further cancer research

CONTACTS AND LOCATIONS:
Locations (1):
- Mackay Memorial Hospital, Taipei, Zhongshan Dist, Taiwan